CLINICAL TRIAL: NCT03690414
Title: A One-month, Randomized, Single Centre, Double-masked, Comparative Study to Evaluate the Short-term Ocular Effects of Experimental BHVI2 and 0.02% Atropine Eye Drops Either Alone or in Combination
Brief Title: Evaluation of Short Term Use of Experimental Eye Drops BHVI2, 0.02% Atropine and BHVI2 Plus 0.02% Atropine Eye Drops
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hai Yen Eye Care (Industry)
Collaborators: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VCRTC-2018-01
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-02

CONDITIONS: Myopia
Keywords: Myopia control; Atropine eye drops; Caffeine eye drops; Pupillary diameter; Accommodative responses
MeSH Terms: conditions — Myopia | interventions — Atropine; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Children aged between 6 to 13 years old. Myopia with spherical equivalent of -0.50D or worse with cylinder of -2.00D or less
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study treatments will be labelled as A, B and C at the Pharmacy. The masked study products will then be sent to the study coordinator to dispense
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental BHVI2 eye drops (Active Comparator): 20 participants will receive one drop per eye every night for four weeks.
  Interventions: Drug: Experimental BHVI2
- 0.02% Atropine eye drops (Active Comparator): 20 participants will receive one drop per eye every night for four weeks.
  Interventions: Drug: Atropine sulfate 0.02% eye drops
- Experimental BHVI2 plus 0.02% atropine (Active Comparator): 20 participants will receive one drop per eye every night for four weeks.
  Interventions: Combination Product: Combination eye drops

INTERVENTIONS:
Drug: Experimental BHVI2 — Experimental BHVI2 eye drops
  Arms: Experimental BHVI2 eye drops
Drug: Atropine sulfate 0.02% eye drops — Atropine eye drops
  Arms: 0.02% Atropine eye drops
Combination Product: Combination eye drops — Combination eye drops with experimental BHVI2 plus 0.02% atropine
  Arms: Experimental BHVI2 plus 0.02% atropine

SUMMARY:
To assess the one-month ocular effects of nightly application of experimental BHVI2 and 0.02% atropine eye drops either alone or in combination, in children aged between 6 to 13 years old with myopia and randomized to use of experimental BHVI2 eye drops, 0.02% atropine eye drops, experimental BHVI2 plus 0.02% atropine eye drops.

DETAILED DESCRIPTION:
Atropine was proven to be effective in controlling myopia. 7-methylxanthine was considered to play a role in slowing myopia. The experimental BHVI2 eye drops were proven to be safe for in-eye use in the trial that was conducted in Sydney, Australia. The investigators wish to evaluate the effects of experimental BHVI2 and 0.02% atropine eye drops either alone or in combination mainly on the pupillary and accommodative responses in children aged between 6 to 13 years old over a one-month period.

ELIGIBILITY:
Inclusion Criteria:

* be accompanied by a parent or guardian who is able to read and comprehend Vietnamese/English and give informed consent as demonstrated by signing a record of informed consent;
* at baseline, be within the age range of 6 to 13 years old inclusive;
* be diagnosed as myopic having spherical equivalent between -0.50 diopter and-6.00 diopter.
* willing to comply with the applying eye drops once nightly at bedtime and follow the clinical trial visit schedule as directed by the Investigator.
* be willing to comply with the wearing and clinical trial visit schedule as directed by the investigator;
* have ocular findings deemed to be normal
* vision correctable to at least 20/25 or better in each eye with spectacles

Exclusion Criteria:

Subjects enrolled in the trial must NOT have:

* Any pre-existing ocular irritation, allergic conjunctivitis, injury or condition, including infection or disease.
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants.
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial.
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial.
* NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used.
* History of eye trauma
* History of use of myopia control interventions such as Orthokeratology or eye surgery.
* Contraindications to atropine and caffeine such as pulmonary disease, heart conditions and ADHD
* Known allergy or intolerance to ingredients to atropine eye-drops, xanthines and other derivatives of anti-muscarinic receptor agents.
* Currently enrolled in another clinical trial.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in pupillary diameter | At baseline, at two-week and one-month visits
  Measure and compare the photopic and mesopic pupil size (milimeters) before and after instillation of eye drops
Change in accommodative amplitude | At baseline, at two-week and one-month visits
  Measure and compare the accommodative amplitude (diopters) before and after instillation of eye drops

CONTACTS AND LOCATIONS:
Overall Officials: Huy D.M Tran, MD, MSc, Principal Investigator — Hai Eye Eye Care
Locations (1):
- Department of Ophthalmology - An Sinh Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Bruce A. Re: Holden et al.: Global prevalence of myopia and high myopia and temporal trends from 2000 through 2050 (Ophthalmology 2016;123:1036-1042). Ophthalmology. 2017 Mar;124(3):e24-e25. doi: 10.1016/j.ophtha.2016.06.066. No abstract available. PMID 28219507
- [Background] Sankaridurg PR, Holden BA. Practical applications to modify and control the development of ametropia. Eye (Lond). 2014 Feb;28(2):134-41. doi: 10.1038/eye.2013.255. Epub 2013 Dec 6. PMID 24310242
- [Background] Huang J, Wen D, Wang Q, McAlinden C, Flitcroft I, Chen H, Saw SM, Chen H, Bao F, Zhao Y, Hu L, Li X, Gao R, Lu W, Du Y, Jinag Z, Yu A, Lian H, Jiang Q, Yu Y, Qu J. Efficacy Comparison of 16 Interventions for Myopia Control in Children: A Network Meta-analysis. Ophthalmology. 2016 Apr;123(4):697-708. doi: 10.1016/j.ophtha.2015.11.010. Epub 2016 Jan 27. PMID 26826749
- [Background] Shih YF, Chen CH, Chou AC, Ho TC, Lin LL, Hung PT. Effects of different concentrations of atropine on controlling myopia in myopic children. J Ocul Pharmacol Ther. 1999 Feb;15(1):85-90. doi: 10.1089/jop.1999.15.85. PMID 10048351
- [Background] Clark TY, Clark RA. Atropine 0.01% Eyedrops Significantly Reduce the Progression of Childhood Myopia. J Ocul Pharmacol Ther. 2015 Nov;31(9):541-5. doi: 10.1089/jop.2015.0043. Epub 2015 Jul 28. PMID 26218150
- [Background] Chatzistefanou KI, Mills MD. The role of drug treatment in children with strabismus and amblyopia. Paediatr Drugs. 2000 Mar-Apr;2(2):91-100. doi: 10.2165/00148581-200002020-00002. PMID 10937461
- [Background] Chen AM, Cotter SA. The Amblyopia Treatment Studies: Implications for Clinical Practice. Adv Ophthalmol Optom. 2016 Aug;1(1):287-305. doi: 10.1016/j.yaoo.2016.03.007. No abstract available. PMID 28435934
- [Background] Chia A, Lu QS, Tan D. Five-Year Clinical Trial on Atropine for the Treatment of Myopia 2: Myopia Control with Atropine 0.01% Eyedrops. Ophthalmology. 2016 Feb;123(2):391-399. doi: 10.1016/j.ophtha.2015.07.004. Epub 2015 Aug 11. PMID 26271839
- [Background] Tran HDM, Tran YH, Tran TD, Jong M, Coroneo M, Sankaridurg P. A Review of Myopia Control with Atropine. J Ocul Pharmacol Ther. 2018 Jun;34(5):374-379. doi: 10.1089/jop.2017.0144. Epub 2018 May 1. PMID 29715053
- [Background] Shih KC, Chan TC, Ng AL, Lai JS, Li WW, Cheng AC, Fan DS. Use of Atropine for Prevention of Childhood Myopia Progression in Clinical Practice. Eye Contact Lens. 2016 Jan;42(1):16-23. doi: 10.1097/ICL.0000000000000189. PMID 26340385
- [Background] Chia A, Chua WH, Cheung YB, Wong WL, Lingham A, Fong A, Tan D. Atropine for the treatment of childhood myopia: safety and efficacy of 0.5%, 0.1%, and 0.01% doses (Atropine for the Treatment of Myopia 2). Ophthalmology. 2012 Feb;119(2):347-54. doi: 10.1016/j.ophtha.2011.07.031. Epub 2011 Oct 2. PMID 21963266
- [Background] Chia A, Chua WH, Wen L, Fong A, Goon YY, Tan D. Atropine for the treatment of childhood myopia: changes after stopping atropine 0.01%, 0.1% and 0.5%. Am J Ophthalmol. 2014 Feb;157(2):451-457.e1. doi: 10.1016/j.ajo.2013.09.020. Epub 2013 Dec 4. PMID 24315293
- [Background] Chua WH, Balakrishnan V, Chan YH, Tong L, Ling Y, Quah BL, Tan D. Atropine for the treatment of childhood myopia. Ophthalmology. 2006 Dec;113(12):2285-91. doi: 10.1016/j.ophtha.2006.05.062. Epub 2006 Sep 25. PMID 16996612
- [Background] Shih YF, Hsiao CK, Chen CJ, Chang CW, Hung PT, Lin LL. An intervention trial on efficacy of atropine and multi-focal glasses in controlling myopic progression. Acta Ophthalmol Scand. 2001 Jun;79(3):233-6. doi: 10.1034/j.1600-0420.2001.790304.x. PMID 11401629
- [Background] North RV, Kelly ME. A review of the uses and adverse effects of topical administration of atropine. Ophthalmic Physiol Opt. 1987;7(2):109-14. doi: 10.1111/j.1475-1313.1987.tb01004.x. PMID 2958765
- [Background] Kennedy RH, Dyer JA, Kennedy MA, Parulkar S, Kurland LT, Herman DC, McIntire D, Jacobs D, Luepker RV. Reducing the progression of myopia with atropine: a long term cohort study of Olmsted County students. Binocul Vis Strabismus Q. 2000;15(3 Suppl):281-304. PMID 11486796
- [Background] Syniuta LA, Isenberg SJ. Atropine and bifocals can slow the progression of myopia in children. Binocul Vis Strabismus Q. 2001;16(3):203-8. PMID 11511287
- [Background] Wu PC, Yang YH, Fang PC. The long-term results of using low-concentration atropine eye drops for controlling myopia progression in schoolchildren. J Ocul Pharmacol Ther. 2011 Oct;27(5):461-6. doi: 10.1089/jop.2011.0027. Epub 2011 Aug 4. PMID 21815829